CLINICAL TRIAL: NCT07339007
Title: Observational Study to Validate a Family Physician Echocardiography Training Programme
Acronym: HEART-CAMFiC
Status: Enrolling by invitation | Type: Observational
Sponsor: Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Collaborators: University of Barcelona (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Monica Solanes Cabus, Vice President, Societat Catalana de Medicina Familiar i Comunitaria (CAMFiC), Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC)
Other Study IDs: HEART-CAMFiC FoCUS Study Group
Record Dates: First submitted 2025-12-10; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Valvular Heart Diseases; Atrial Fibrillation (AF); Arterial Hypertension; Cardiomyopathies
Keywords: Primary Health Care; Echocardiography; Family Practice; Ultrasound Training; Ultrasonography; Education, Medical
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases; Atrial Fibrillation; Hypertension; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort of GPs: Cohort of GPs:
  Board-certified Family and Community Medicine specialists in Catalonia who will complete a structured FoCUS training programme and participate in a validation study.
  Intervention of interest: FoCUS training (online theory + supervised hands-on practice, including simulator assessment) followed by routine FoCUS use in primary care with data capture in REDCap and paired comparison with cardiologist echocardiography.
  Inclusion criteria: Family and Community Medicine specialist; CAMFiC member; workplace access to an ultrasound device suitable for FoCUS; commitment to complete the programme.
  Exclusion criteria: Not meeting any inclusion criterion.
  Interventions: Other: Cohort of GPs: Training program
- Cohort of Patients: Cohort of Patients:
  Individuals aged >18 years who require cardiac imaging for any clinical indication in routine care at a site where a participating GP works.
  Intervention of interest: A FoCUS assessment performed by the trained GP as part of usual clinical care; no additional study tests or follow-up visits.
  Sampling: Non-random, consecutive/clinician-driven recruitment based on routine clinical need and medical judgment.
  Exclusion criteria: Refusal to participate (no written informed consent) and severe mental illness or significant cognitive impairment preventing informed consent.
  Interventions: Diagnostic Test: Cohort of patients

INTERVENTIONS:
Other: Cohort of GPs: Training program — 1. Accredited curriculum: 18 hours of online theory (2.7 CCFCPS credits) with a mandatory 20-item MCQ assessing knowledge and image interpretation.
  2. Structured, supervised scanning volume: 4-hour hands-on introductory session on core cardiac views using healthy volunteers, followed by 70 hours of supervised clinical training with a hospital cardiologist, including a predefinied target of 60 FoCUS examinations per GP.
  Groups: Cohort of GPs
Diagnostic Test: Cohort of patients — Eligible patients are those seen in routine primary care by participating GPs who, based on usual clinical judgment, need an echocardiographic assessment. In these cases, the GP will perform a FoCUS scan as part of the consultation and record a standard set of variables in the study eCRF. When the patient subsequently undergoes a comprehensive echocardiography in cardiology, both assessments (GP FoCUS and cardiology echocardiography) will be paired to evaluate agreement. No additional tests or extra study visits are required beyond usual care.
  Groups: Cohort of Patients

SUMMARY:
Observational Study on the Validation of Family Doctors' Training in Echocardiography

The Catalan Society of Family and Community Medicine (CAMFiC) developed a structured training program for Family Physicians in focused cardiac ultrasound (FoCUS). This study evaluates GP FoCUS performance against comprehensive echocardiography and assesses training competence.

Developed between September 2023 and November 2025 (92 hours total, including 70 hours supervised practice), participants perform FoCUS on patients with suspected cardiac pathology. The study measures concordance between GP FoCUS and cardiologist echocardiography, and evaluates FoCUS integration into primary care pathways to enhance diagnostic capacity for common cardiac conditions.

DETAILED DESCRIPTION:
ACKGROUND & JUSTIFICATION Cardiovascular disease generates long cardiology waiting lists in Spain (>90 days echocardiography). Elderly patients discharged from hospital require cardiac follow-up in primary care, but Family Medicine residency (MIR) excludes point-of-care ultrasound (POCUS) training. This gap limits GP triage capacity for common cardiac pathology.

The Catalan Society of Family and Community Medicine (CAMFiC), in collaboration with the Catalan Society of Cardiology (SCC), developed a structured FoCUS training program (2022, 92 hours total: 18h theory + 4h workshop for cardiac views + 70h supervised hospital practice) to empower primary care physicians.

HYPOTHESIS

Primary Hypotheses:

1. Structured FoCUS training enables GPs to achieve competency across ≥6/7 predefined domains (standard views, LVEF estimation, RV/volume assessment, valvular disease detection, pericardial effusion, LVH recognition, theoretical knowledge).
2. This training program achieves ≥80% concordance between GP-performed FoCUS and cardiologist-performed standard echocardiography on predefined cardiac parameters (κ≥0.6).

   Secondary Hypotheses:
3. Trained GP will be able to integrate this technique into routine practice (≥1 scan/week).
4. FoCUS enables documentation of key cardiac pathologies (LVEF impairment, RV dilation, significant valve disease, pericardial effusion) among primary care scans performed for clinical indications (dyspnea, heart murmur, suspected HF, arrhythmia).
5. FoCUS plus clinical data identifies ≥3 distinct patient profiles among primary care patients assessed.
6. FoCUS in primary care achieves appropriate triage of patients requiring formal echocardiography.
7. The programme will be acceptable to stakeholders, with high satisfaction reported by patients, family doctors, and cardiologists participating in the programme.
8. FoCUS in primary care will increase identification of suspected heart failure among assessed patients and may reduce time to appropriate management.

STUDY OVERVIEW Prospective observational study (CEIm IDIAP 23/072-P). 46 CAMFiC GPs perform FoCUS on consecutive adult patients (>18 years) with clinical cardiac indication during primary care visits, followed by cardiologist echocardiography confirmation. Data captured via REDCap eCRF.

See Outcomes, Eligibility Criteria, and Arms/Interventions for specific measures, criteria, and procedures.

PHASES

* Phase 0: Preparation (2022)
* Phase 1: Training (2022-2025)
* Phase 2: Data collection (2024-2027)
* Phase 3: Analysis (kappa/ICC/Bland-Altman, mixed models) (2027-2028)
* Phase 4: Dissemination (PhD thesis, peer-reviewed publications) (2028)

CLINICAL IMPACT Reduces time-to-diagnosis, shortens cardiology waiting lists, enables primary care triage of common cardiac conditions, cost-effective, scalable model.

PROTOCOL AVAILABILITY Full protocol available upon request from IDIAP Jordi Gol Primary Care Research Institute.

See structured sections (Outcomes, Eligibility Criteria, Arms/Interventions) for specific measures, criteria, and procedures.

ELIGIBILITY:
* Inclusion/Exclusion Criteria for Professionals:

Inclusion criteria for professionals in the training program are:

* Board-certified specialist in Family and Community Medicine.
* Member of the Catalan Society of Family and Community Medicine (CAMFiC).
* Access at the workplace to an ultrasound device suitable for FoCUS.
* Willing and able to complete all training and study procedures. Exclusion criteria: Not meeting any inclusion criterion.

  * Inclusion/Exclusion Criteria for Patients:

The inclusion criteria for patients are:

* Age over 18 years old.
* Clinical indication for FoCUS/echocardiographic assessment in routine care.
* Attended at a site where a participating GP provides care.
* Able to provide written informed consent.

Exclusion criteria:

* Refusal to participate (no written informed consent)
* Severe mental illness
* Significant cognitive impairment preventing informed consent.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of:
  * GPs who meet the eligibility criteria and complete the FoCUS training programme, regardless of workplace setting.
  * Patients aged >15 years receiving routine care at sites where participating GPs work, in whom a FoCUS assessment is clinically indicated, and who provide written informed consent for inclusion in the paired FoCUS-comprehensive echocardiography agreemnt study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between GP-performed FoCUS and cardiologist-performed standard echocardiography. | Diagnostic agreement assessment in real-world clinical practice following training completion (2024-2027 recruitment period).
  Agreement between GP-performed FoCUS and cardiologist-performed standard echocardiography on key cardiac parameters: left ventricular systolic function (preserved vs. reduced), cavity sizes (normal vs. dilated), and significant valve abnormalities (none vs. moderate-severe). Additional parameters include pericardial effusion and IVC dilation. Measured by weighted kappa coefficient comparing blinded independent interpretations of the same patients. Higher κ = better agreement. Clinical competency threshold κ ≥ 0.6 (substantial agreement).
  Unit of measure: Weighted kappa coefficient (0-1)

SECONDARY OUTCOMES:
GPs knowledge and competence after FoCUS training | Training completion (6-8 months post-enrolment)
  Change from baseline in 20-item MCQ knowledge score + % practical competencies checklist + simulator pass rate, assessing FoCUS training effectiveness for GPs (Objective 1).
FoCUS routine integration in clinical practice | Following completion of recruitment (December 2027), a survey will be conducted among the 46 family physicians who have participated in this training program to assess the proportion regularly applying FoCUS (≥1/week) in routine primary care consultation
  Proportion of trained GPs regularly using FoCUS (≥1/week) in primary care consultations, assessed by participant survey at end of recruitment (Objective 3).
FoCUS indications and abnormalities documented. | Documentation analysis of FoCUS performed during study period for clinical indications and documented key abnormalities: first half of 2028 (January-June 2028), following recruitment completion and REDCap data extraction.
  Frequency of predefined indications (dyspnea, heart murmur, suspected heart failure, cardiac arrhythmia) and key abnormalities documented during routine FoCUS use (Objective 4).
Time from FoCUS triage to specialist care | Real-world implementation (2024-2027)
  Time elapsed from the detection of significant cardiac findings using FoCUS to care by a specialist/echocardiography in general practitioners trained in FoCUS versus standard care, evaluating the benefits of triage and accelerated care pathways (hypothesis 6+8).
Programme acceptability and satisfaction | Programme completion (2027)
  Satisfaction scores (1-5 Likert scale) from patients, GPs, and cardiologists regarding FoCUS programme acceptability and usability (Objective 7).

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sisó-Almirall, Ph.D., Study Director — IDIBAPS. CAMFiC.; Laura Conangla-Ferrín, Ph.D., Study Director — Institut Catlà de la Salut. CAMFiC
Locations (1):
- Societat Catalana de Medicina Familiar i Comunitària (CAMFiC), Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Patient data will be collected in a pseudonymised format in REDCap, a secure platform for clinical research data management. Access to the dataset will be restricted to authorised members of the research team and used solely to address the study objectives. Data handling will comply with applicable data protection regulations, safeguarding confidentiality throughout the study and subsequent analyses. There is no plan to share individual participant data (IPD) outside the study team.

REFERENCES:
- [Background] Solanes-Cabús M, Pujol-Salud J, Alonso-Aliaga J, Mayench-Ariza F, Marsal-Mora JR, Sabaté-Navarro A, et al. Inter-rater agreement and reliability among general practitioners and radiologists on ultrasound examinations after a specialized training program [Internet]. Journal of Primary Health Care & General Practice. 2019;3(1):026 [cited 2025 Oct 25]. Available from: https://www.scribd.com/document/877574246/
- [Background] Sorensen B, Hunskaar S. Point-of-care ultrasound in primary care: a systematic review of generalist performed point-of-care ultrasound in unselected populations. Ultrasound J. 2019 Nov 19;11(1):31. doi: 10.1186/s13089-019-0145-4. PMID 31749019
- [Background] British Medical Ultrasound Society; Royal College of Radiologists. Recommendations for specialists practising ultrasound independently of radiology departments: safety, governance and education [Internet]. London: Royal College of Radiologists; 2023 Apr [cited 2025 Oct 26]. Available from: https://www.rcr.ac.uk/publication/recommendations-for-specialists-practising-ultrasound-independently-of-radiology-departments-safety-governance-and-education/
- [Background] Conangla-Ferrin L, Guirado-Vila P, Solanes-Cabus M, Teixido-Gimeno D, Diez-Garcia L, Pujol-Salud J, Evangelista-Robleda L, Bertran-Culla J, Ortega-Vila Y, Canal-Casals V, Siso-Almirall A. Ultrasound in primary care: Consensus recommendations on its applications and training. Results of a 3-round Delphi study. Eur J Gen Pract. 2022 Dec;28(1):253-259. doi: 10.1080/13814788.2022.2150163. PMID 36503353
- [Background] Homar V, Gale ZK, Lainscak M, Svab I. Knowledge and skills required to perform point-of-care ultrasonography in family practice - a modified Delphi study among family physicians in Slovenia. BMC Fam Pract. 2020 Mar 26;21(1):56. doi: 10.1186/s12875-020-01130-z. PMID 32216753
- [Background] Diaz-Gomez JL, Mayo PH, Koenig SJ. Point-of-Care Ultrasonography. N Engl J Med. 2021 Oct 21;385(17):1593-1602. doi: 10.1056/NEJMra1916062. No abstract available. PMID 34670045
- [Background] Andersen CA, Lundbye-Christensen S, Riis A, Mehnert U, Lokkegaard T, Mengel-Jorgensen T, Rasmussen LD, Soll N, Stork B, Andersen SK, Pil L, Stjernebjerg C, Graumann O, Jensen MB. General practitioners' scanning competence following tailored ultrasound training: a hybrid effectiveness-implementation study. BMC Med Educ. 2025 May 20;25(1):733. doi: 10.1186/s12909-025-07356-8. PMID 40394656
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. BMJ. 2007 Oct 20;335(7624):806-8. doi: 10.1136/bmj.39335.541782.AD. PMID 17947786
- [Background] Cascos E, Sitges M. The inevitable lightness of echocardioscopy: teamwork, training and quality assurance are indispensable. Rev Esp Cardiol (Engl Ed). 2023 Feb;76(2):83-85. doi: 10.1016/j.rec.2022.09.003. Epub 2022 Sep 19. No abstract available. English, Spanish. PMID 36245100
- [Background] Evangelista Robleda L. Utilidad de la ecoscopia realizada por un médico de familia en el diagnóstico de la enfermedad cardiovascular en atención primaria [doctoral thesis]. Barcelona: Universidad Autónoma de Barcelona; 2015. Available at: https://ddd.uab.cat/pub/tesis/2015/hdl_10803_328411/ler1de1.pdf
- [Background] Bult MM, van de Ree TF, Wind AM, Hurley KM, van de Ree MA. The use of echocardiography compared to electrocardiogram when screening for left ventricular hypertrophy in hypertensive patients: A cross-sectional study. J Clin Hypertens (Greenwich). 2024 Aug;26(8):977-985. doi: 10.1111/jch.14867. Epub 2024 Jul 4. PMID 38963706
- [Background] Cheng S, He J, Han Y, Han S, Li P, Liao H, Guo J. Global burden of atrial fibrillation/atrial flutter and its attributable risk factors from 1990 to 2021. Europace. 2024 Jul 2;26(7):euae195. doi: 10.1093/europace/euae195. PMID 38984719
- [Background] Camm CF, Von Ende A, Gajendragadkar PR, Pessoa-Amorim G, Mafham M, Allen N, Parish S, Casadei B, Hopewell JC. Role of primary and secondary care data in atrial fibrillation ascertainment: impact on risk factor associations, patient management, and mortality in UK Biobank. Europace. 2025 Feb 5;27(2):euae291. doi: 10.1093/europace/euae291. PMID 39910980
- [Background] World Health Organization. Global burden of stroke [Internet]. [accessed 30-07-2024]. Available at: https://www.emro.who.int/health-topics/stroke-cerebrovascular-accident/index.html
- [Background] King's College London, for the Stroke Alliance for Europe. The burden of stroke in Europe. Atrial fibrillation [Internet]. [consultat 1 gener 2024].
- [Background] Cameli M, Mandoli GE, Ambrosio G, Cerbai E, Coiro S, Emdin M, Marcucci R, Morrone D, Palazzuoli A, Savino K, Padeletti L, Mondillo S, Pedrinelli R; Societa Italiana di Cardiologia, Sezione Regionale Tosco-Umbra. Arterial hypertension and atrial fibrillation: standard and advanced echocardiography from diagnosis to prognostication. J Cardiovasc Med (Hagerstown). 2018 Feb;19(2):51-61. doi: 10.2459/JCM.0000000000000607. PMID 29251696
- [Background] d'Arcy JL, Coffey S, Loudon MA, Kennedy A, Pearson-Stuttard J, Birks J, Frangou E, Farmer AJ, Mant D, Wilson J, Myerson SG, Prendergast BD. Large-scale community echocardiographic screening reveals a major burden of undiagnosed valvular heart disease in older people: the OxVALVE Population Cohort Study. Eur Heart J. 2016 Dec 14;37(47):3515-3522. doi: 10.1093/eurheartj/ehw229. Epub 2016 Jun 26. PMID 27354049
- [Background] Williams C, Mateescu A, Rees E, Truman K, Elliott C, Bahlay B, Wallis A, Ionescu A. Point-of-care echocardiographic screening for left-sided valve heart disease: high yield and affordable cost in an elderly cohort recruited in primary practice. Echo Res Pract. 2019 Jul 16;6(3):71-79. doi: 10.1530/ERP-19-0011. eCollection 2019 Sep. PMID 31475072
- [Background] Thoenes M, Bramlage P, Zamorano P, Messika-Zeitoun D, Wendt D, Kasel M, Kurucova J, Steeds RP. Patient screening for early detection of aortic stenosis (AS)-review of current practice and future perspectives. J Thorac Dis. 2018 Sep;10(9):5584-5594. doi: 10.21037/jtd.2018.09.02. PMID 30416809
- [Background] Potter A, Pearce K, Hilmy N. The benefits of echocardiography in primary care. Br J Gen Pract. 2019 Jul;69(684):358-359. doi: 10.3399/bjgp19X704513. No abstract available. PMID 31249096
- [Background] Davidsen AH, Andersen S, Halvorsen PA, Schirmer H, Reierth E, Melbye H. Diagnostic accuracy of heart auscultation for detecting valve disease: a systematic review. BMJ Open. 2023 Mar 24;13(3):e068121. doi: 10.1136/bmjopen-2022-068121. PMID 36963797
- [Background] Gardezi SKM, Myerson SG, Chambers J, Coffey S, d'Arcy J, Hobbs FDR, Holt J, Kennedy A, Loudon M, Prendergast A, Prothero A, Wilson J, Prendergast BD. Cardiac auscultation poorly predicts the presence of valvular heart disease in asymptomatic primary care patients. Heart. 2018 Nov;104(22):1832-1835. doi: 10.1136/heartjnl-2018-313082. Epub 2018 May 24. PMID 29794244
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, et al. 2021 ESC/EACTS Guidelines for the management of valvular heart disease: developed by the Task Force of the European Society of Cardiology and the European Association for Cardio-Thoracic Surgery. Eur Heart J. 2022;43(7):561-632. doi:10.1093/eurheartj/ehab395.
- [Background] Anderson K, Ross HJ, Austin PC, Fang J, Lee DS. Health Care Use Before First Heart Failure Hospitalization: Identifying Opportunities to Pre-Emptively Diagnose Impending Decompensation. JACC Heart Fail. 2020 Dec;8(12):1024-1034. doi: 10.1016/j.jchf.2020.07.008. Epub 2020 Nov 11. PMID 33189631
- [Background] Abdin A, Anker SD, Butler J, Coats AJS, Kindermann I, Lainscak M, Lund LH, Metra M, Mullens W, Rosano G, Slawik J, Wintrich J, Bohm M. 'Time is prognosis' in heart failure: time-to-treatment initiation as a modifiable risk factor. ESC Heart Fail. 2021 Dec;8(6):4444-4453. doi: 10.1002/ehf2.13646. Epub 2021 Oct 16. PMID 34655282
- [Background] Panisello-Tafalla A, Haro-Montoya M, Caballol-Angelats R, Montelongo-Sol M, Rodriguez-Carralero Y, Lucas-Noll J, Clua-Espuny JL. Prognostic Significance of Lung Ultrasound for Heart Failure Patient Management in Primary Care: A Systematic Review. J Clin Med. 2024 Apr 23;13(9):2460. doi: 10.3390/jcm13092460. PMID 38730988
- [Background] Conangla-Ferrin L. Validez de la ecografía pulmonar en el diagnóstico de la insuficiencia cardiaca en atención primaria [doctoral thesis]. Barcelona: Universitat Autònoma de Barcelona; 2024.
- [Background] Maestre A, Gallego J, Aznar J, Mora A, Martín-Hidalgo A. Precisión diagnóstica de los criterios clínicos para identificar la insuficiencia cardíaca sistólica y diastólica: estudio transversal. Rev Eval Práct Clin. 2017;15(1):55-6.
- [Background] Cohen SS, Roger VL, Weston SA, Jiang R, Movva N, Yusuf AA, Chamberlain AM. Evaluation of claims-based computable phenotypes to identify heart failure patients with preserved ejection fraction. Pharmacol Res Perspect. 2020 Dec;8(6):e00676. doi: 10.1002/prp2.676. PMID 33124771
- [Background] Koudstaal S, Pujades-Rodriguez M, Denaxas S, Gho JMIH, Shah AD, Yu N, Patel RS, Gale CP, Hoes AW, Cleland JG, Asselbergs FW, Hemingway H. Prognostic burden of heart failure recorded in primary care, acute hospital admissions, or both: a population-based linked electronic health record cohort study in 2.1 million people. Eur J Heart Fail. 2017 Sep;19(9):1119-1127. doi: 10.1002/ejhf.709. Epub 2016 Dec 23. PMID 28008698
- [Background] Bachtiger P, Kelshiker MA, Petri CF, Gandhi M, Shah M, Kamalati T, Khan SA, Hooper G, Stephens J, Alrumayh A, Barton C, Kramer DB, Plymen CM, Peters NS. Survival and health economic outcomes in heart failure diagnosed at hospital admission versus community settings: a propensity-matched analysis. BMJ Health Care Inform. 2023 Mar;30(1):e100718. doi: 10.1136/bmjhci-2022-100718. PMID 36921978
- [Background] Heidenreich P, Sandhu A. Advances in management of heart failure. BMJ. 2024;385.
- [Background] Anguita-Sanchez M, Crespo-Leiro MG, de Teresa-Galván E, Jiménez-Navarro M, Alonso-Pulpón L, Muñiz-García J. Prevalencia de la insuficiencia cardiaca en la población general española mayor de 45 años. Estudio PRICE. Rev Esp Cardiol. 2008;61(10):1041-9.
- [Background] Canadian Point of Care Ultrasound Society. Courses - POCUS Education [Internet]. Canada: CPOCUS; [consultat 03-03-2025]. Available at: https://cpocus.ca/
- [Background] European Association of Cardiovascular Imaging. Focus e-learning course [Internet]. European Society of Cardiology; [accessed 03-03-2025]. Available at: https://www.escardio.org/Sub-specialty-communities/European-Association-of-Cardiovascular-Imaging-(EACVI)/Education/focus-e-learning-course
- [Background] Chaptal M, Tendron L, Claret PG, Muller L, Markarian T, Mattatia L, Roger C, de la Coussaye JE, Pelaccia T, Bobbia X. Focused Cardiac Ultrasound: A Prospective Randomized Study of Simulator-Based Training. J Am Soc Echocardiogr. 2020 Mar;33(3):404-406. doi: 10.1016/j.echo.2019.10.010. Epub 2019 Dec 19. No abstract available. PMID 31864772
- [Background] Mackay FD, Zhou F, Lewis D, Fraser J, Atkinson PR. Can You Teach Yourself Point-of-care Ultrasound to a Level of Clinical Competency? Evaluation of a Self-directed Simulation-based Training Program. Cureus. 2018 Sep 17;10(9):e3320. doi: 10.7759/cureus.3320. PMID 30473953
- [Background] Bowcock EM, Morris IS, Mclean AS, Orde SR. Basic critical care echocardiography: How many studies equate to competence? A pilot study using high fidelity echocardiography simulation. J Intensive Care Soc. 2017 Aug;18(3):198-205. doi: 10.1177/1751143717700166. Epub 2017 Apr 18. PMID 29118831
- [Background] Neskovic AN, Skinner H, Price S, Via G, De Hert S, Stankovic I, Galderisi M, Donal E, Muraru D, Sloth E, Gargani L, Cardim N, Stefanidis A, Cameli M, Habib G, Cosyns B, Lancellotti P, Edvardsen T, Popescu BA; Reviewers: This document was reviewed by members of the 2016-2018 EACVI Scientific Documents Committee. Focus cardiac ultrasound core curriculum and core syllabus of the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2018 May 1;19(5):475-481. doi: 10.1093/ehjci/jey006. PMID 29529170
- [Background] Olesen LL, Andersen A, Thaulow S. Hand-held echocardiography is useful for diagnosis of left systolic dysfunction in an elderly population. Dan Med J. 2015 Jul;62(7):A5100. PMID 26183043
- [Background] Hammadah M, Ponce C, Sorajja P, Cavalcante JL, Garcia S, Gossl M. Point-of-care ultrasound: Closing guideline gaps in screening for valvular heart disease. Clin Cardiol. 2020 Dec;43(12):1368-1375. doi: 10.1002/clc.23499. Epub 2020 Nov 11. PMID 33174635
- [Background] Kovell LC, Ali MT, Hays AG, Metkus TS, Madrazo JA, Corretti MC, Mayer SA, Abraham TP, Shapiro EP, Mukherjee M. Defining the Role of Point-of-Care Ultrasound in Cardiovascular Disease. Am J Cardiol. 2018 Oct 15;122(8):1443-1450. doi: 10.1016/j.amjcard.2018.06.054. Epub 2018 Jul 19. PMID 30115421
- [Background] Doherty JU, Kort S, Mehran R, Schoenhagen P, Soman P; Rating Panel Members; Appropriate Use Criteria Task Force. ACC/AATS/AHA/ASE/ASNC/HRS/SCAI/SCCT/SCMR/STS 2019 Appropriate Use Criteria for Multimodality Imaging in the Assessment of Cardiac Structure and Function in Nonvalvular Heart Disease : A Report of the American College of Cardiology Appropriate Use Criteria Task Force, American Association for Thoracic Surgery, American Heart Association, American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, and the Society of Thoracic Surgeons. J Nucl Cardiol. 2019 Aug;26(4):1392-1413. doi: 10.1007/s12350-019-01751-7. PMID 31250324
- [Background] Waweru-Siika W, Pluddemann A, Heneghan C. Focused Cardiac Ultrasound Training for Non-cardiologists: An Overview and Recommendations for a Lower Middle-Income Country. Crit Care Clin. 2022 Oct;38(4):827-837. doi: 10.1016/j.ccc.2022.06.015. PMID 36162913
- [Background] Kirkpatrick JN, Grimm R, Johri AM, Kimura BJ, Kort S, Labovitz AJ, Lanspa M, Phillip S, Raza S, Thorson K, Turner J. Recommendations for Echocardiography Laboratories Participating in Cardiac Point of Care Cardiac Ultrasound (POCUS) and Critical Care Echocardiography Training: Report from the American Society of Echocardiography. J Am Soc Echocardiogr. 2020 Apr;33(4):409-422.e4. doi: 10.1016/j.echo.2020.01.008. Epub 2020 Feb 29. No abstract available. PMID 32122742
- [Background] Johri AM, Durbin J, Newbigging J, Tanzola R, Chow R, De S, Tam J. Cardiac Point-of-Care Ultrasound: State-of-the-Art in Medical School Education. J Am Soc Echocardiogr. 2018 Jul;31(7):749-760. doi: 10.1016/j.echo.2018.01.014. Epub 2018 Mar 15. PMID 29550326
- [Background] Jujo S, Lee-Jayaram JJ, Sakka BI, Nakahira A, Kataoka A, Izumo M, Kusunose K, Athinartrattanapong N, Oikawa S, Berg BW. Pre-clinical medical student cardiac point-of-care ultrasound curriculum based on the American Society of Echocardiography recommendations: a pilot and feasibility study. Pilot Feasibility Stud. 2021 Sep 14;7(1):175. doi: 10.1186/s40814-021-00910-3. PMID 34521479
- [Background] Pérez de Isla L, Díaz Sánchez S, Pagola J, Garcia de Casasola G, López Fernández T, Sánchez Barrancos IM, et al. Documento de consenso de SEMI, semFYC, SEN y SEC sobre ecocardioscopia en España. Rev Esp Cardiol. 2018;71(11):883-90.
- [Background] Chugh Y, Lohese O, Sorajja P, Garberich R, Stanberry L, Cavalcante J, Gossl M. Adoptability and accuracy of point-of-care ultrasound in screening for valvular heart disease in the primary care setting. J Clin Ultrasound. 2022 Feb;50(2):265-270. doi: 10.1002/jcu.23062. Epub 2021 Sep 7. PMID 34818437
- [Background] Morbach C, Buck T, Rost C, Peter S, Gunther S, Stork S, Prettin C, Erbel R, Ertl G, Angermann CE; Handheld-BNP Research Network. Point-of-care B-type natriuretic peptide and portable echocardiography for assessment of patients with suspected heart failure in primary care: rationale and design of the three-part Handheld-BNP program and results of the training study. Clin Res Cardiol. 2018 Feb;107(2):95-107. doi: 10.1007/s00392-017-1181-3. Epub 2017 Nov 15. PMID 29143161
- [Background] Evangelista A, Galuppo V, Mendez J, Evangelista L, Arpal L, Rubio C, Vergara M, Liceran M, Lopez F, Sales C, Miralles V, Galinsoga A, Perez J, Arteaga M, Salvador B, Lopez C, Garcia-Dorado D. Hand-held cardiac ultrasound screening performed by family doctors with remote expert support interpretation. Heart. 2016 Mar;102(5):376-82. doi: 10.1136/heartjnl-2015-308421. Epub 2016 Jan 22. PMID 26802099
- [Background] Luong CL, Ong K, Kaila K, Pellikka PA, Gin K, Tsang TSM. Focused Cardiac Ultrasonography: Current Applications and Future Directions. J Ultrasound Med. 2019 Apr;38(4):865-876. doi: 10.1002/jum.14773. Epub 2018 Aug 26. PMID 30146784
- [Background] Spencer KT, Flachskampf FA. Focused Cardiac Ultrasonography. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1243-1253. doi: 10.1016/j.jcmg.2018.12.036. PMID 31272607
- [Background] Barron KR, Wagner MS, Hunt PS, Rao VV, Bell FE, Abdel-Ghani S, Schrift D, Norton D, Bornemann PH, Haddad R, Hoppmann RA. A Primary Care Ultrasound Fellowship: Training for Clinical Practice and Future Educators. J Ultrasound Med. 2019 Apr;38(4):1061-1068. doi: 10.1002/jum.14772. Epub 2018 Sep 4. PMID 30182369
- [Background] Andersen CA, Holden S, Vela J, Rathleff MS, Jensen MB. Point-of-Care Ultrasound in General Practice: A Systematic Review. Ann Fam Med. 2019 Jan;17(1):61-69. doi: 10.1370/afm.2330. PMID 30670398
- [Background] Esquerra M, Roura Poch P, Masat Tico T, Canal V, Maideu Mir J, Cruxent R. [Abdominal ultrasound: a diagnostic tool within the reach of general practitioners]. Aten Primaria. 2012 Oct;44(10):576-83. doi: 10.1016/j.aprim.2011.07.016. Epub 2011 Oct 22. Spanish. PMID 22018792
- [Background] Programa formativo de la especialidad de Medicina Familiar y Comunitaria. Ministerio de Sanidad y Consumo. 7188. BOE num. 105. Orden SCO/1198/2005, de 3 de marzo, por la que se aprueba y publica el programa formativo de la especialidad de Medicina Familiar y Comunitaria. https://www.boe.es/buscar/doc.php?id=BOE-A-2005-7188
- [Background] Indicadores clínicos en Atención Primaria. Factores de riesgo y enfermedad cardiovascular. Ministerio de Sanidad, Consumo y Bienestar Social. 01/02/2019. https://www.sanidad.gob.es/estadEstudios/estadisticas/estadisticas/estMinisterio/SIAP /BDCAP_Indic_clinic_Cardiovasc_2016.pdf
- [Background] Introducció de l'ecografia clínica a l'atenció́ primària i comunitària. Departament de Salut. Generalitat de Catalunya. Febrer 2022. https://salutweb.gencat.cat/web/.content/_departament/ambits-estrategics/atencio- primaria-comunitaria/docs/introduccio-ecografia-clinica-apic.pdf